CLINICAL TRIAL: NCT07375472
Title: he Effect of Virtual Reality Headset, Squishy (Squeeze Toy), and Poetry Reading on Postoperative Pain Control After Total Knee Arthroplasty
Brief Title: Distraction Techniques for Postoperative Pain After Total Knee Arthroplasty: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Tinaztepe University (Other)
Responsible Party: Principal Investigator, Berna Dizer, Assistant professor, Izmir Tinaztepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: İzmirTınaztepeÜ-B.Dizer-003
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Total Knee Arthroplasty; Postoperative Pain
Keywords: virtual reality; distraction technique; postoperative pain; total knee arthroplasty; nursing intervention
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Virtual Reality (VR) Headset (Experimental): Participants will receive routine postoperative care and standard analgesia according to the hospital protocol. In addition, they will receive a structured distraction intervention using a virtual reality (VR) headset during the postoperative pain period while hospitalized (e.g., within the first 24 hours after surgery). The VR content is delivered under supervision at the bedside as a non-pharmacological distraction method.
  Interventions: Behavioral: VR Distraction
- Squishy (Squeeze Toy) (Experimental): Participants will receive routine postoperative care and standard analgesia according to the hospital protocol. In addition, they will use a squishy (squeeze toy) as a tactile distraction method during the postoperative pain period while hospitalized (e.g., within the first 24 hours after surgery). Participants are instructed to use the squeeze toy during episodes of pain/discomfort as a non-pharmacological distraction technique.
  Interventions: Behavioral: Tactile Distraction With Squishy
- Poetry Reading (Experimental): Participants will receive routine postoperative care and standard analgesia according to the hospital protocol. In addition, they will perform poetry reading as a cognitive distraction method during the postoperative pain period while hospitalized (e.g., within the first 24 hours after surgery). Poetry reading is provided as a structured non-pharmacological distraction intervention at the bedside.
  Interventions: Behavioral: Poetry Reading Distraction
- Usual Care Control (No Intervention): articipants will receive routine postoperative care and standard analgesia according to the hospital protocol. No structured distraction intervention (VR, squishy, or poetry reading) will be provided.

INTERVENTIONS:
Behavioral: VR Distraction — A supervised virtual reality distraction session delivered via a VR headset during postoperative hospitalization to support non-pharmacological pain management.
  Other Names: Virtual Reality (VR) Headset Distraction
  Arms: Virtual Reality (VR) Headset
Behavioral: Tactile Distraction With Squishy — Use of a squishy (squeeze toy) as a tactile distraction technique during postoperative hospitalization as part of non-pharmacological pain management.
  Other Names: Squeeze Toy (Squishy) Distraction
  Arms: Squishy (Squeeze Toy)
Behavioral: Poetry Reading Distraction — Structured poetry reading conducted during postoperative hospitalization as a cognitive distraction approach to support non-pharmacological pain management.
  Other Names: Poetry Reading
  Arms: Poetry Reading

SUMMARY:
This randomized controlled trial evaluates the effectiveness of three distraction techniques-virtual reality (VR) headset, squishy (squeeze toy), and poetry reading-on postoperative pain control in adults undergoing total knee arthroplasty. Participants are randomized into four parallel groups (three intervention arms and one usual care control). Pain intensity is assessed using the Visual Analog Scale (VAS), with primary assessment at 24 hours after surgery.

DETAILED DESCRIPTION:
Total knee arthroplasty is a common orthopedic procedure that can be associated with significant postoperative pain. In addition to standard pharmacological analgesia, non-pharmacological approaches such as distraction techniques may help reduce perceived pain by redirecting attention away from nociceptive stimuli. This single-center, parallel-group randomized controlled trial will be conducted in the Orthopedics and Traumatology Clinic of Osmaniye State Hospital in Türkiye. Eligible adults (≥18 years) undergoing total knee arthroplasty will be randomized using a stratified block randomization approach based on baseline pain severity (VAS 0-3, 4-6, 7-10) to ensure balanced allocation across groups. The intervention arms include (1) VR headset distraction, (2) use of a squishy (squeeze toy) as a tactile distraction method, and (3) poetry reading as a cognitive distraction method. The control group receives usual postoperative care without a structured distraction intervention. All groups follow the same postoperative analgesia protocol. The primary outcome is postoperative pain intensity measured by VAS at 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Undergoing total knee arthroplasty
* Hospitalized in the postoperative period at Osmaniye State Hospital
* Able to communicate and complete pain assessment (Visual Analog Scale)
* Provides written informed consent
* Managed under the same postoperative analgesia protocol and operated by the same surgeon (as per study protocol)

Exclusion Criteria:

* Severe cognitive impairment or inability to provide valid pain assessment
* Postoperative complications that may interfere with participation or pain assessment
* Contraindication to the assigned distraction method (e.g., intolerance to wearing a VR headset, severe nausea/dizziness, claustrophobia)
* Refusal or withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (VAS) | 24 hours after surgery
  Visual Analog Scale pain score (0=no pain, 10=worst pain).

SECONDARY OUTCOMES:
Pain Intensity (VAS) by Pain Severity Strata | 24 hours after surgery
  VAS pain score analyzed by baseline pain strata (0-3, 4-6, 7-10) using stratified allocation groups.

CONTACTS AND LOCATIONS:
Overall Officials: Songül Gungor, Principal Investigator — Osmaniye State Hospital; Berna Dizer, Study Director — Izmir Tinaztepe University
Locations (1):
- Osmaniye State Hospital, Osmaniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The informed consent/IRB approval did not include permission for public deposition of individual participant-level data. In accordance with local privacy regulations in Türkiye (e.g., KVKK), individual participant data will not be shared publicly. De-identified and aggregated data may be provided by the corresponding author upon reasonable request under a data-use agreement.